CLINICAL TRIAL: NCT05539807
Title: Short and Long-term Changes in Eating Disorder Symptoms During and After a Low-threshold Mindfulness-based Intervention Administered by a Self-help Organization in Norway
Brief Title: Mindfulness and Eating Disorder Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Ingrid Dundas, Associate Professor, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK353216
Record Dates: First submitted 2022-08-24; First posted 2022-09-14 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Eating Disorders
Keywords: Eating Disorder; Mindfulness; Self-compassion; Longitudinal; Within-person; Long-term
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All participants receive the intervention
  Interventions: Behavioral: Mindful Eating Conscious Living

INTERVENTIONS:
Behavioral: Mindful Eating Conscious Living — MECL is a 8 week mindfulness-based group intervention. Each session is of 2.5-3 hours duration. During the sessions, theories about eating-related difficulties in general are presented, participants are guided in mindfulness practices and participants who want to share their experiences in the group can do so. Topics include: (1) What is mindfulness, why and how can we use mindfulness in relation to eating (2) slowing down, taking breaks and noticing different types of "hunger" (e.g. physical hunger and the "hunger" for comfort - "heart hunger) (3) working with satiety and satisfaction (4) becoming aware of patterns associated with one's eating behaviors, (5) awareness of feelings and bodily sensations (6) Food and mood (7) craving, and finally (8) working with "heart hunger" and emotional eating. Six to 10 participants participated in each group.

SUMMARY:
This prospective one-arm study aims to examine short and long-term changes in dysfunctional eating among individuals who signed up for an 8-week, group based, low threshold, mindfulness-based intervention. The study is an extension of a quality assurance project which was provided by a nation-wide self-help organization for people with self-identified eating problems. Eating disorder symptoms and the proposed predictors (self-kindness, self-judgment and mindfulness) were registered online at 12 measurement time points. In the current study we will invite the same participants to complete the same measures four years after the intervention.

DETAILED DESCRIPTION:
Recent literature-reviews suggest that mindfulness-based interventions may be effective in treating problems related to dysfunctional eating such as binge eating and emotional eating. Less is known about the processes through which change happens. Moreover, long-term follow-up is scarce. The main aim of the current project is to examine the role of self-kindness and self-judgement in predicting changes in eating disorder symptoms four years after, and to analyze longitudinal data for the entire project. Measures were administrated before the intervention, each week during the intervention, after the intervention, at follow-up 6 months after the intervention and at a second follow up four years after the intervention.

The intervention is an 8-week mindfulness-based eating program (Mindful Eating Conscious Living). This intervention was administered by a nation-wide Norwegian self-help eating disorder organization. Participants who enrolled in the program (N=197) were asked to complete standardized self-report instruments at recruitment (T1), digitally during each of the 8-week sessions (T2-T9), after the intervention was completed (T10) and six months after the intervention was completed (T11).

The current study - a PhD project - will invite the same participants to complete the same measures four years after completing the program. This will provide a rich data set, collected over four years.

The main hypotheses are:

Self-kindness and self-judgment as predictors of ED symptoms

1. During the intervention, self-kindness and self-judgment at a given week will predict eating disorder (ED) symptoms the following week (within-person).
2. Level of self-kindness and self-judgement will predict the level of ED symptoms during the whole course (pre, each week during the intervention, post and four-year follow-up) (between-person).

3) Pre-post changes in self-kindness and self-judgment will predict level of ED symptoms at six-month and four-year follow up (between-person changes)

Secondary hypotheses are:

4) During the intervention, mindfulness (from the self-compassion scale) at a given week will predict ED symptoms the following week (within-person change) 5) Level of mindfulness will predict the level of ED symptoms during the whole course (pre, each week during the intervention, post and four-year follow-up) (between-person).

6) Pre-post changes in mindfulness and mindful eating will predict changes in ED symptoms, and relationship and life-satisfaction, at six month and four-year follow-up (between-person changes).

7) Pre-post changes in shame will predict changes in ED symptoms at six month and four-year follow-up (between-person change).

8) During the intervention, expectations for positive effects of the intervention, will predict ED symptoms at the next week (within-person change).

9) Who the instructor is, will predict pre-post changes in outcome. For each within-person hypothesis, the reverse effects will also be examined.

Qualitative part of study:

A randomly selected sub-group of 20 participants will be interviewed about their experiences during and after the intervention.

Statistical Analysis Plan These longitudinal data will be disaggregated so that within- and between-person effects can be studied separately Repeated measurements like the present one typically has drop-outs and missing data. Therefore, we will use mixed models instead of paired t-tests, repeated measures ANOVAs, and ordinary linear regression to analyze the data. Mixed models use maximum likelihood estimation, which is the state-of-the-art approach to handle missing data (Schafer & Graham, 2002). Especially if data are missing at random, which is likely in our study, mixed models give more unbiased results than the other analytic methods.

In preliminary analyses, and for each of the dependent variables (EDE-Q, subscales form Self-compassion Scale), the combination of random effects and covariance structure of residuals that gives the best fit for the "empty" model (the model without fixed predictors except the intercept) will be chosen. Akaike's Information Criterion (AIC) will be used to compare the fit of different models. Models that give a reduction in AIC greater than 2 will be considered better (Burnham & Anderson, 2004). The program SPSS version 28.0.1.1 (15) will be used.

Possible transformations:

All variables will be assessed in their original and validated format as is recommended practice, as long as this is possible with regards to statistical assumptions underlying the pre-defined analyses (i.e., multiple regression). However, if this is not possible with regards to the statistical assumptions behind the analyses, transformation (e.g., square root or log-transformations) may be needed to apply interval-based methods. The investigators will examine the degree of skewness and evaluate this against the assumptions and analyses before choosing the appropriate analysis. The pre-registered and planned analyses include multiple regression as long as assumptions are met. Alternatively, a non-parametric test will be used.

Inference criteria:

We pre-define the significance level: p < 0.05 to determine significance.

Missing data:

Maximum likelihood

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as having a binge-eating related problem and being 16 years or older.

Exclusion Criteria:

* High suicidal risk, serious self-harm, active psychosis, active major depressive episode, anorexia nervosa, BMI < 18, or debilitating social anxiety.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Change in eating disorder symptoms measured by Eating Disorder Examination Questionnaire (EDE-Q) | Pre, weekly during treatment - 8 weeks, post, 6 months follow-up, four years follow-up
  A self-report questionnaire measuring eating disorder symptoms by Fairburn and colleagues
Change in self-kindness, self-judgement and mindfulness from the Self-compassion scale | Pre, weekly during treatment - 8 weeks, post, 6 months follow-up, four years follow-up
  Subscales from the self-compassion scale of Kristin Neff and colleagues. Self-kindness indicates the tendency to respond with kindness to own feelings of distress and failure (e.g. I try to be understanding and patient towards those aspects of my personality I don't like). Self-judgment indicates the tendency to respond with self-judgment to own feelings of distress and failure (self-judgment, e.g. I'm disapproving and judgmental about my own flaws and inadequacies). Mindfulness indicates the tendency to respond with balanced awareness to own feelings of distress and failure. E.g.: "When something painful happens I try to take a balanced view of the situation".

SECONDARY OUTCOMES:
Change in mindful eating as measured by the Mindful Eating Questionnaire | Pre, post, 6 months follow up, four-years follow-up
  A self-report questionnaire developed by Framson et al asking respondents to indicate the extent to which they engage in mindful eating, e.g. with a nonjudgmental awareness of physical and emotional sensations associated with eating. Sample item: "I notice when there are subtle flavors in the foods I eat".
Change in relationship and life Satisfaction | Pre, post, 6 months follow up, four-years follow-up
  Four items from the Norwegian directory of health's "minimum subjective check list"

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Dundas, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Deidentified quantitative data will be shared.
Time Frame: After completion of the study and for five years.
Access Criteria: Data will be deposited in relevant data depositories and shared with researchers with legitimate interest who's research seems ethically sound.